CLINICAL TRIAL: NCT07036263
Title: "Effect of Oculomotor Therapy in Individuals With Convergence Insufficiency: A Blind Randomized Clinical Trial"
Brief Title: Effect of Oculomotor Therapy in Individuals With Convergence Insufficiency
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Fabiano Politti, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CI-2025
Record Dates: First submitted 2025-06-12; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Convergence Insufficiency
Keywords: Convergence insufficiency; Postural control; Clinical trial
MeSH Terms: conditions — Ocular Motility Disorders

STUDY DESIGN:
Intervention Model Description: Assignment randomised clinical trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (EG) (Experimental): This group will receive treatment with oculomotor therapy
  Interventions: Other: Oculomotor therapy
- Control group (CG) (Other): This group will not receive any type of treatment
  Interventions: Other: No Treatment Added

INTERVENTIONS:
Other: Oculomotor therapy — Oculomotor therapy will follow and adapt the protocol for treating convergence insufficiency (CI). Procedures will be organized progressively, from easiest to most difficult. Gross convergence techniques: (1) Brock String: A 1.5-2 m cord with colored beads; the patient focuses on each bead to train binocular fusion, observing the "X" shape of the cord. (2) Barillé Chart: A card with paired images for each eye; the patient merges the images into one using convergence and sensory fusion. Accommodative techniques: (1) Eccentric Circles: Printed circles with eccentric marks; viewed through filters to train motor and sensory fusion by aligning them into a single 3D image. (2) Opaque Lifesaver Cards: Cards with figures on an opaque background, used with red-green filters to stimulate convergence and fixation by reducing peripheral stimuli and enhancing visual attention.
  Arms: Experimental Group (EG)
Other: No Treatment Added — Participants in the control group will not receive any type of treatment for a period of five weeks. After this period, they will be re-evaluated
  Arms: Control group (CG)

SUMMARY:
The aim of this study is to investigate the effect of oculomotor therapy in individuals with ocular convergence insufficiency.

DETAILED DESCRIPTION:
Seventy participants with convergence insufficiency (CI) will be randomly allocated into two groups: Experimental Group (EG) (n=35) and Control Group (CG) (n=35). The primary outcome will be CI assessed by the convergence test. Secondary outcomes will include quality of life, postural balance, and gait speed. The EG will undergo five sessions of oculomotor therapy (once a week), based on and adapted from the established protocol for CI treatment. Results: Outcomes will be assessed by blinded evaluators at baseline, one week after the end of the treatment, and at 1 and 3 months follow-up. The CG will not receive any intervention. Data will be analyzed using statistical tests with a significance level set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with convergence insufficiency (CI);
* Aged between 18 and 60 years;
* Physically active individuals;
* Without cognitive impairments;
* Without vestibular system impairments (e.g., dizziness).

Exclusion Criteria:

* Diagnosis of neurodegenerative diseases (e.g., Parkinson's, ALS);
* Presence of dementia;
* History of stroke;
* Presence of vestibular disorders;
* Systemic neuromuscular diseases;
* Disabling musculoskeletal pain;
* Diagnosis of diabetic polyneuropathy;
* Use of joint prostheses;
* Ongoing physical therapy treatment;
* Lack of physical ability to perform the prescribed physical activities.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
General mobility | 3 months
  General mobility will be assessed using the Timed 'Up-and-Go' test with time measured in seconds as the unit of measurement.

SECONDARY OUTCOMES:
Single-Leg Stance Test | 3 months
  The single-leg stance test is used to assess static balance and predict frailty, particularly in community-dwelling older adults. Participants will be asked to stand on one leg for a maximum of 30 seconds, first with eyes open and then with eyes closed. The duration will be measured in three trials per visual condition, and the longest time will be considered. Longer stance duration indicates better balance. The examiner will remain beside the participant to prevent any risk of falling.
Postural Control Assessment | 3 months
  Postural control will be evaluated using a force platform (BIOMEC 400 v1.1, EMG System Ltda®). Tests will be performed under four conditions: (1) eyes open; (2) eyes closed; (3) eyes open, single-leg stance (dominant leg); and (4) eyes closed, single-leg stance (dominant leg). The main parameters will be the center of pressure (CoP) sway velocity (cm/s), in both anteroposterior (AP) and mediolateral (ML) directions.

IPD SHARING:
Plan to Share IPD: No